CLINICAL TRIAL: NCT03443921
Title: Artery Divestment Technique in Artery-Involved Pancreatic Cancer: A Single-Institution, Open-Labeled Randomized Controlled Trial
Brief Title: Divestment for Artery-involved Pancreatic Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Yi Miao, Director of Pancreas Center, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMU-JSPH-PC-DIV
Record Dates: First submitted 2017-12-17; First posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Pancreatic Cancer; Locally Advanced Pancreatic Cancer; Neoadjuvant Therapy; Borderline Resectable Pancreatic Cancer
Keywords: Artery Divestment Technique; Locally Advanced Pancreatic Cancer; Neoadjuvant Therapy; Borderline Resectable Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery Group (Experimental): In Surgery Group, an artery divestment combined pancreatectomy will be performed if no pre-operative contra-indication or intra-operative metastasis were revealed. Post-operative adjuvant chemotherapies were prescribed according to performance status.
  Interventions: Procedure: Artery Divestment Technique
- NeoChemo Group (Active Comparator): In NeoChemo (Neoadjuvant Chemotherapy) Group, neoadjuvant chemotherapy will be utilized. After 2 circles of neoadjuvant chemotherapies, patients will be reevaluated and curative operation would be attempted if without disease progression.
  Interventions: Drug: Nab-paclitaxel

INTERVENTIONS:
Procedure: Artery Divestment Technique — Tunica adventitia was pick up by forceps and opened by electrocoagulation at 1 cm distal from tumor-artery contact. Space between tunica adventitia and external elastic lamina (EEL) were blunt lifting tumor-invaded adventitia by angled clamp. Adventitia was then sectioned to show EEL. Loose dissect space could be achieve along long the plane between EEL and adventitia as long as tumor invasion outside EEL. Tumor and invaded adventitia were further cut open by electrocoagulation proximally. Circumferentially, separation could be done by blunt dissection around EEL. Nourishing blood vessels of the artery would be secured by electrocoagulation or ultrasonic scalpel while major branch would be ligated or transfixed.
  Other Names: Sub-adventitial Resection
  Arms: Surgery Group
Drug: Nab-paclitaxel — After eligibility testing as blood tests, contrast-enhanced CT and MRI scan, 3 cycles were administered (1,000 mg/m2 of gemcitabine and 125 mg/m2 of nab-paclitaxel on days 1, 8, and 15 every 28 days).Patients will be reevaluated and curative operation would be attempted if without disease progression.
  Arms: NeoChemo Group

SUMMARY:
Pancreatic cancer is the most lethal malignancy of human being. Surgery is the only potential cure of pancreatic cancer. The invasion of major abdominal arteries is one of the most important factor restricting surgical intervention. For artery-involved pancreatic cancer (ai-PC) patients, pre-operative adjuvant therapies, especially the neoadjuvant chemotherapy, has brought exciting postoperative survival. Yet due to the potential screening effect of this treatment strategy, nearly half of ai-PC patients failed to benefit from surgery because of disease progression, adverse reactions of adjuvant treatment and other reasons. Artery divestment for the treatment of ai-PC firstly reported by our center, can significantly increase resection rate and produce overall survival benefit in some patients. This study is to explore whether up-front surgery with artery divestment combined curative pancreatectomy or the chemotherapy-first strategy would be more beneficial for ai-PC patients' survival.

Subjects will be randomized to treatment group either receiving up-front artery divestment combined pancreatectomy (Surgery Group) or adjuvant chemotherapies (Chemo Group). In Surgery Group, an artery divestment combined pancreatectomy will be performed if no pre-operative contra-indication or intra-operative metastasis were revealed. Post-operative adjuvant chemotherapies were prescribed according to performance status. In Chemo Group, adjuvant chemotherapy of gemcitabine or gemcitabine + cisplatin will be utilized according to performance status. After 2 circles of adjuvant chemotherapies, patients will be reevaluated and curative operation would be attempted if without disease progression.

Overall mortality at one year after randomization will be the primary endpoint. Other parameters as overall survival after 2 and 3 years, median survival, disease-free survival, margin status of subjects receiving curative surgery, etc. will also be observed.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with pancreatic cancer staged at cT4NxM0(AJCC Cancer Staging Manual, 8th Edition) based on contrast enhanced CT&MRI scan and tumor markers;
2. Age > 18 year and <80 year;
3. Agree to participate in the study with signed informed consent.

Exclusion Criteria:

1. Evidence of metastasis based on physical examination, enhanced CT or enhanced MRI;
2. Poor performance status and/or co-morbidity precluding pancreatectomy and chemotherapy;
3. Focal vessel narrowing or contour irregularity revealed by radiology examinations;
4. Economic situations cannot afford designed treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Overall mortality at one year after randomization; | 1 year

SECONDARY OUTCOMES:
Overall survival rate after 2 years from randomization; | 2 years
Overall survival rate after 3 years from randomization; | 3 years
Median survival | 3 years
Disease-free survival | 3 years
Margin status of subjects receiving curative surgery | 1 years
  The margin status will be reported as R0, R1 and R2 according to AJCC Cancer Staging Manual 8th ed.
Intra-operative blood transfusion | 1 years
  For both Surgery Group and participants who received operations in NeoChemo Group, category and volume of intra-operative blood transfusion will be reported.
Intra-operative blood loss | 1 years
  For both Surgery Group and participants who received operations in NeoChemo Group, intra-operative blood loss will be measured and reported by milliliter.
Overall surgical complication rate | 1 years
  Overall surgical complication rate for both Surgery Group and participants who received operations in NeoChemo Group will be reported. Post-operative pancreatic fistula, delayed gastric emptying, post-operative hemorrhage, Surgical site infection and other surgical complications will be recorded. Percentage that candidates suffered from surgical complications of surgical cases for both group will be reported.
Incidence of post-operative pancreatic fistula | 1 years
  Post-operative pancreatic fistula (POPF) will be accessed byInternational Study Group of Pancreatic Surgery (ISGPS) standards; Incidence of post-operative pancreatic fistula of surgical cases in both group will be reported.
Incidence of delayed gastric emptying | 1 years
  Delayed gastric emptying (DGE) will be accessed byInternational Study Group of Pancreatic Surgery (ISGPS) standards; Incidence of DGE of surgical cases in both group will be reported.
Incidence of post-operative hemorrhage | 1 years
  Post-operative hemorrhage (POH) will be accessed byInternational Study Group of Pancreatic Surgery (ISGPS) standards; Incidence of POH of surgical cases in both group will be reported.
Incidence of surgical site infection | 1 years
  Surgical site infection was assessed as US CDC guidelines.Incidence of surgical site infection of surgical cases in both group will be reported.
Incidence of other surgical complications | 1 years
  Any other undesirable situations that considered complicated with surgery will be recorded. Incidence of other surgical complications of surgical cases in both group will be reported.
Severe adverse events rate | 3 years
  Feasibility of chemotherapy will be evaluated according to Common Terminology Criteria for Adverse Events, US NCI. Participants receiving neo-adjuvant, adjuvant or palliative chemotherapy will be accessed. Grade 3-5 adverse events, dose reduction or dose delay will be reported.
Quality of life at 0.5 year after randomization | 0.5 year
  EORTC QLQ-C30 (V3.0) will be enrolled to evaluate quality of life.
Quality of life at 1 year after randomization | 1 year
  EORTC QLQ-C30 (V3.0) will be enrolled to evaluate quality of life.
Quality of life at 2 years after randomization | 2 years
  EORTC QLQ-C30 (V3.0) will be enrolled to evaluate quality of life.
Quality of life at 3 years after randomization | 3 years
  EORTC QLQ-C30 (V3.0) will be enrolled to evaluate quality of life.
Performance status at 0.5 year after randomization | 0.5 year
  Karnofsky Performance Status Scale will be enrolled to evaluate Performance status.
Performance status at 1 year after randomization | 1 year
  Karnofsky Performance Status Scale will be enrolled to evaluate Performance status.
Performance status at 2 years after randomization | 2 years
  Karnofsky Performance Status Scale will be enrolled to evaluate Performance status.
Performance status at 3 years after randomization | 3 years
  Karnofsky Performance Status Scale will be enrolled to evaluate Performance status.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Ryan DP, Hong TS, Bardeesy N. Pancreatic adenocarcinoma. N Engl J Med. 2014 Nov 27;371(22):2140-1. doi: 10.1056/NEJMc1412266. No abstract available. PMID 25427123
- [Background] Zhang H, Wroblewski K, Jiang Y, Penney BC, Appelbaum D, Simon CA, Salgia R, Pu Y. A new PET/CT volumetric prognostic index for non-small cell lung cancer. Lung Cancer. 2015 Jul;89(1):43-9. doi: 10.1016/j.lungcan.2015.03.023. Epub 2015 Apr 9. PMID 25936471
- [Background] Tang K, Lu W, Qin W, Wu Y. Neoadjuvant therapy for patients with borderline resectable pancreatic cancer: A systematic review and meta-analysis of response and resection percentages. Pancreatology. 2016 Jan-Feb;16(1):28-37. doi: 10.1016/j.pan.2015.11.007. Epub 2015 Dec 2. PMID 26687001
- [Background] Siegel RL, Miller KD, Jemal A. Cancer Statistics, 2017. CA Cancer J Clin. 2017 Jan;67(1):7-30. doi: 10.3322/caac.21387. Epub 2017 Jan 5. PMID 28055103
- [Background] Seufferlein T, Bachet JB, Van Cutsem E, Rougier P; ESMO Guidelines Working Group. Pancreatic adenocarcinoma: ESMO-ESDO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2012 Oct;23 Suppl 7:vii33-40. doi: 10.1093/annonc/mds224. No abstract available. PMID 22997452
- [Background] Fortner JG, Kim DK, Cubilla A, Turnbull A, Pahnke LD, Shils ME. Regional pancreatectomy: en bloc pancreatic, portal vein and lymph node resection. Ann Surg. 1977 Jul;186(1):42-50. doi: 10.1097/00000658-197707000-00007. PMID 195543
- [Background] Chua TC, Saxena A. Extended pancreaticoduodenectomy with vascular resection for pancreatic cancer: a systematic review. J Gastrointest Surg. 2010 Sep;14(9):1442-52. doi: 10.1007/s11605-009-1129-7. Epub 2010 Apr 9. PMID 20379794